CLINICAL TRIAL: NCT07033663
Title: Study of the Impact of Intrauterine Exposure to Immunomodulatory Drugs on the Development of the Immune System of Children Born to Mothers With Chronic Inflammatory or Oncologic Diseases: The NEWborn-IMM-PACT Study
Brief Title: Impact of In Utero Exposure to Immunomodulatory Drugs on Neonatal Immune System Development
Acronym: NEWbornIMMPACT
Status: Recruiting | Type: Observational
Sponsor: Fundació Sant Joan de Déu (Other)
Collaborators: Hospital Clinic of Barcelona (Other); Hospital Vall d'Hebron (Other)
Responsible Party: Sponsor
Other Study IDs: NEWborn-IMM-PACT
Record Dates: First submitted 2025-05-28; First posted 2025-06-24 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-05

CONDITIONS: Pregnancy Related; Immune-mediated Diseases
Keywords: monoclonal antibodies; pregnancy; immunomodulators
MeSH Terms: interventions — Antibodies, Monoclonal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples Without DNA — Serum, plasma, PBMCs, RNA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pregnant women with chronic inflammatory and/or oncological diseases exposed to mAb during pregnancy: Study Population:
  Inclusion criteria: Pregnant women with immune-mediated inflammatory or oncologic diseases, categorized into:
  1. High-exposed group: IMD treatment throughout pregnancy.
  2. Low-exposed group: IMD treatment limited to the first/second trimester.
  3. Non-exposed group: No IMD exposure or treatment with non-placental-crossing biologics, serving as a control to distinguish immunological changes attributable to maternal disease.
  Newborns and an age- and sex-matched healthy control group (0-12 months) will be included.
  Exclusion criteria for mother and child: lack of signed informed consent, primary immunodeficiencies, active infection at the time of sampling or significant comorbidities.
  Interventions: Drug: Monoclonal antibody

INTERVENTIONS:
Drug: Monoclonal antibody — non-intervention. Drug used in clinical practice as per practitioner decision
  Other Names: non-intervention. Drug used in clinical practice

SUMMARY:
What is this project about? This project aims to better understand how the immune system develops in babies whose mothers received immunomodulatory treatments during pregnancy. These treatments are necessary for women with autoimmune, inflammatory, allergic, or cancer-related diseases who cannot stop their medication while pregnant.

Why is it important? Although these treatments help keep the mother and baby healthy, some medications can cross the placenta and affect the baby's immune system. Since pregnant women are usually not included in clinical trials, the investigators still don't know exactly how these drugs might influence the baby's immune development.

How will the investigators do it? The investigators will follow a group of pregnant women receiving these treatments and monitor their babies at birth, and at 3, 6, and 12 months. The study will take place in three leading hospitals in Spain: Hospital Sant Joan de Déu, Hospital Clínic, and Vall d'Hebron. The investigators will also use organoid models in the lab to better understand how these drugs affect fetal development.

Who will benefit? This study will help parents concerned about the impact of treatments during pregnancy on their child's health. It will also give doctors the evidence they need to make safer treatment decisions, and support the creation of new clinical guidelines to protect both mothers and babies.

DETAILED DESCRIPTION:
The use of immunomodulatory drugs (IMD) in chronic inflammatory or oncologic diseases is increasingly widespread in pregnant women who have gestational desire and need to keep their disease under control for the safety of pregnancy. General objective: analyze the safety of IMD exposure during pregnancy used in clinical practice on the development of the newborn immune system. Specific objectives: 1) To evaluate lymphoid organogenesis, including regulatory T/B populations, and the direct effect on the drug target immune pathway, in cord and peripheral blood of newborns exposed in utero to biologic immunomodulators (bIMD, monoclonals and fusion protein); 2) To evaluate the epigenetic fingerprint in cord and peripheral blood of newborns exposed in utero to bIMD; 3) To develop an in vitro model (organoid-platform) to study the impact of IMD and maternal disease in the fetal period. 4) To develop a guide of specific recommendations, which includes the perspective of the newborn. Methods: Observational multicenter prospective cohort study of infants exposed to bIMD during pregnancy, born to mothers with chronic inflammatory or oncologic diseases. Clinical and analytical follow-up, from birth, at 3,6 and 12 months. Clinical: general health status, data on infections or autoimmune or allergic events. Analytical: serum levels of bIMD, maturation and function of T and B extended lymphocyte populations, integrity of the bIMD target pathway, study of epigenetic changes. The results will be compared with a control population. In vitro study: organoid-based models obtained from hiPSCs differentiated towards hematopoietic components; B-cell maturation will be evaluated after different IMD exposure. The investigators expect to: 1) surmount the knowledge gap on the impact of in utero IMD exposure, to define the newborn infectious risk, of autoimmunity and/or allergy, and 2) to be create and disseminate protocols of follow-up specific to them.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women with immune-mediated inflammatory or oncologic diseases, categorized into:

1. High-exposed group: monoclonal treatment throughout pregnancy.
2. Low-exposed group: monoclonal treatment limited to the first/second trimester.
3. Non-exposed group: No monoclonal exposure or treatment with non-placental-crossing biologics, serving as a control to distinguish immunological changes attributable to maternal disease.

   -

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women with immune-mediated inflammatory or oncologic diseases. 90 mother-child pairs: 15 per each of the 6 disease groups: rheumatology, neuroimmunology, dermatology, inflammatory bowel disease, allergy, and oncology.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Growth | first 12 months of age
  Growth will be measured with OMS scale. The World Health Organization (WHO) Child Growth Standards (0-5 years) and WHO Growth Reference (5-19 years) use Z-scores to assess growth, typically ranging from -6 to +6, with most values between -3 and +3. Higher scores indicate greater body size, which can mean better growth (e.g., height-for-age) or a worse outcome (e.g., overweight or obesity in BMI-for-age), depending on the growth index used.
Neurodevelopment | first 12 months of age
  Neurodevelopment will be measured with Haizea-Llevant scale. The Haizea-Llevant scale is a standardized tool used in Spain to assess neurodevelopment in children aged 0 to 5 years, based on the Denver Developmental Screening Test. It evaluates development across four domains, and scores are reported as age of acquisition of milestones or percentile ranges, with higher scores indicating better neurodevelopmental outcomes; there is no fixed minimum or maximum, as it depends on age-specific milestones. A child scoring below the 3rd percentile in one or more areas may indicate developmental delay and require further evaluation.
Infection history | first 12 months of age
  Number and type of infections will be recorded
Vaccine response | first 12 months of age
  IgG responses to tetanus, diphtheria and pneumococcus
Hypersensitivity | first 12 months of age
  Atopy, food allergy will be recorded. Atopy and food allergy will be assessed based on clinical history obtained through structured clinical interview and findings from physical examination, following standard diagnostic criteria. No specific questionnaire or scale will be used, as data will be collected descriptively during routine clinical evaluation.
Immune Profiling in neonatal samples: Spectral flow cytometry | first 12 months of age
  Investigators will perform a comprehensive immune cell phenotype (T/B/NK cells, T and B regulatory subsets) from cord and peripheral blood samples and evaluate de % of each cell type to be compared to age-matched healthy controls reference values
Immune Profiling in neonatal samples: T cell function | first 12 months of age
  Investigators will evaluate T cell response to stimulants (PHA, PWM, ConA) and calculate the proliferation capacity in % compared to age-matched healthy controls.
Immune Profiling in neonatal samples: B cell function | first 12 months of age
  Investigators will evaluate B cell function by performing Plasmablast differentiation and measuring immunoglobulin production (IgG, IgA, IgM).
Immune Profiling in neonatal samples: Cytokine profiling | first 12 months of age
  Investigators will perform a 92-cytokine panel (Olink platform, advanced PCR technology) to measure different cytokine abundance in serum samples
Immune Profiling in neonatal samples: IMD Monitoring | first 12 months of age
  Investigators will perform an ELISA-based maternal/neonatal IMD (immunomodulatory drug) concentration analysis to measure drug levels in serum samples
Immune Profiling in neonatal samples: Vaccine responses | first 12 months of age
  Investigators will measure Antibody titers for tetanus, diphtheria, pneumococcus using commercial kits. à afegeix (IgG) despres de antibody titers.

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Hospital Sant Joan de Déu, Esplugues de Llobregat, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebrón, Barcelona